CLINICAL TRIAL: NCT04811755
Title: Is TIme From adMission to surgEry an Independent Prognostic Factor for Survival of Patients With Gastro-intestinal Perforation Associated With Septic Shock: (TIME) An Italian Intersocietary Retrospective and Prospective Observational Trial
Acronym: TIME
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: San Luigi Gonzaga Hospital (Other)
Responsible Party: Principal Investigator, Rossella Reddavid, Doctor, San Luigi Gonzaga Hospital
Other Study IDs: TT.01
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Emergency Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Surgical timing from ED admission to surgery — the impact of delay of time between patient admission to ED and surgery for source control on 90-d mortality and postoperative outcomes in patients with gastrointestinal perforation with or without septic shock

SUMMARY:
Gastro-intestinal perforation is a condition that can become life-threatening in case of appearance of systemic symptoms, sepsis-related peripheral hypoperfusion and single or multiple organ failure needing a prompt intervention in Emergency Department (ED) setting. Literature reports disagreeing data about the effect of surgical timing on mortality and postoperative outcomes: Buck et al. described a 2.4 % of decreased survival every hour of surgical delay in case of perforated peptic ulcers. Other authors documented significantly longer postoperative hospital stay, greater health costs and a significant increase of postoperative complication and mortality rates when surgery is delayed in high-risk patients with comorbidities or age > 65 years. Azuhata described a highly significant relationship between delayed surgery and patients' survival: after 6 hours from admission to ED, patients with gastrointestinal perforation and associated septic shock don't survive to surgery. The aim of this study is to assess the impact of delay of time between patient admission to ED and surgery for source control on 30-d mortality and postoperative outcomes in patients with gastrointestinal perforation with or without septic shock. Furthermore, we want to define the time threshold within which surgery can affect patients' survival.

DETAILED DESCRIPTION:
This is an Italian National multicenter study composed by a retrospective phase of data collection from patients of past ten years and a perspective one of next two years.

INCLUSION AND EXCLUSION CRITERIA We include in our analysis all patients with more than 18 years old undergoing emergency surgery for gastro-intestinal perforations, with or without signs of septic shock. All patients with covered perforations or abdominal perivisceral free air bubbles treated with non- operative management or delayed surgery will be excluded. An online Case Report Form (CRF) will be filled out by every participating Italian participating center.

ENDPOINTS Primary outcome analyzed is in-hospital Clavien-Dindo > 3 complication rate [12]. Secondary outcomes are 60-d mortality rate, total length of stay (LOS), LOS in Intensive Care Unit (ICU), days of mechanical ventilation, re-intervention rate and 30-d readmission rate.

Analyzed variables are:

* Hospital characteristics; teaching/non-teaching setting; I/II level ED; emergency surgery/volume x year; 24H/on-call radiology and surgery team; presence of a dedicated OR in ED;
* Patient demographics (gender, age, Body Mass Index (BMI) and American Society of Anaesthesiologists' (ASA) classification of Physical Health, medical history of past abdominal surgical operations and comorbidities according to Charlson Comorbidity Index (CCI), mainly related to corticosteroids therapy and immunosuppressive conditions),
* Patient management in ED: admission date and time; Priority code at admission; time of abdominal x-Ray; time of CT-scan; Time of patient evaluation by surgeon on- call; Preoperative resuscitation management (Y/N, type, time of beginning); presence of Sepsis (infection documented or suspected + SOFA >=2) and of septic shock (sepsis + persistent hypotension needing vasopressors to maintain a Mean Arterial Pressure (MAP) of 65 mmHg; serum values of lactates > 18 mg/dL (or 2 mmol/L) with an adequate volume resuscitation measures) at admission or during patient stay in ED; SOFA score at admission; Emergency surgery score; ACS NSQIP® Surgical Risk score.
* Radiological findings: CT-scan reports of patients selected will be analyzed by site data-collection centers with the aim to identify typical and atypical radiological findings (subdiaphragmatic free gas, free peritoneal fluid, bowel wall discontinuity, extraluminal oral contrast, extraluminal abscess, abdominal collections, fat stranding, portal venous gas, wall bowel thickening, pneumatosis and mucosal hyperenhancement).
* Surgery: Time of skin incision; Type and duration of surgery; source control surgery, Open Abdomen; surgical approach; site and cause of perforation; pathologic data; Emergency surgery score; ACS NSQIP® Surgical Risk score.
* Postoperative Course: Preoperative mortality (patients die before surgery); Medical and Surgical complications (Clavien-Dindo score); total LOS; LOS in ICU; days of Mechanical Ventilation; Re-intervention rate; 90-d mortality.

PLANNED SAMPLE SIZE With a binary response variable, β=0·95, α=0·05, an anticipated small effect size and an allocation ratio 1:10 (Early treatment Yes vs. No), it has been calculated that 3276 patients are required to detect an association between the variables and the endpoint.

PLANNED ANALYSES Time between patient admission to ED and surgery will be analyzed as a continuous variable with t-Student's tests, comparing means between the different outcomes (primary and secondary). Different cut-off will be tested to define a significant time threshold correlating with outcomes. If necessary, more time intervals will be evaluated to evaluate correlations between the variables collected and the time.

ELIGIBILITY:
Inclusion Criteria:

* more than 18 years old
* emergency surgery for gastro-intestinal perforations
* with or without signs of septic shock

Exclusion Criteria:

* All patients with covered perforations or abdominal perivisceral free air bubbles treated with non- operative management
* delayed surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing emergency surgery for gastro-intestinal perforations, with or without signs of septic shock
Sampling Method: Probability Sample
Enrollment: 3276 (Estimated)
Dates: Start 2009-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
in-hospital Clavien-Dindo > 3 complication rate | up to 90 days after surgery

SECONDARY OUTCOMES:
90-d mortality rate | up to 90 days after surgery
total length of stay (LOS) | up to 90 days after surgery
LOS in Intensive Care Unit (ICU) | up to 90 days after surgery
days of mechanical ventilation | up to 90 days after surgery
re-intervention rate | up to 90 days after surgery
30-d readmission rate | up to 30 days after surgery

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Azuhata T, Kinoshita K, Kawano D, Komatsu T, Sakurai A, Chiba Y, Tanjho K. Time from admission to initiation of surgery for source control is a critical determinant of survival in patients with gastrointestinal perforation with associated septic shock. Crit Care. 2014 May 2;18(3):R87. doi: 10.1186/cc13854. PMID 24886954
- [Result] Buck DL, Vester-Andersen M, Moller MH; Danish Clinical Register of Emergency Surgery. Surgical delay is a critical determinant of survival in perforated peptic ulcer. Br J Surg. 2013 Jul;100(8):1045-9. doi: 10.1002/bjs.9175. PMID 23754645
- [Result] Rhodes A, Evans LE, Alhazzani W, Levy MM, Antonelli M, Ferrer R, Kumar A, Sevransky JE, Sprung CL, Nunnally ME, Rochwerg B, Rubenfeld GD, Angus DC, Annane D, Beale RJ, Bellinghan GJ, Bernard GR, Chiche JD, Coopersmith C, De Backer DP, French CJ, Fujishima S, Gerlach H, Hidalgo JL, Hollenberg SM, Jones AE, Karnad DR, Kleinpell RM, Koh Y, Lisboa TC, Machado FR, Marini JJ, Marshall JC, Mazuski JE, McIntyre LA, McLean AS, Mehta S, Moreno RP, Myburgh J, Navalesi P, Nishida O, Osborn TM, Perner A, Plunkett CM, Ranieri M, Schorr CA, Seckel MA, Seymour CW, Shieh L, Shukri KA, Simpson SQ, Singer M, Thompson BT, Townsend SR, Van der Poll T, Vincent JL, Wiersinga WJ, Zimmerman JL, Dellinger RP. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. Intensive Care Med. 2017 Mar;43(3):304-377. doi: 10.1007/s00134-017-4683-6. Epub 2017 Jan 18. PMID 28101605
- [Result] Sartelli M, Viale P, Catena F, Ansaloni L, Moore E, Malangoni M, Moore FA, Velmahos G, Coimbra R, Ivatury R, Peitzman A, Koike K, Leppaniemi A, Biffl W, Burlew CC, Balogh ZJ, Boffard K, Bendinelli C, Gupta S, Kluger Y, Agresta F, Di Saverio S, Wani I, Escalona A, Ordonez C, Fraga GP, Junior GA, Bala M, Cui Y, Marwah S, Sakakushev B, Kong V, Naidoo N, Ahmed A, Abbas A, Guercioni G, Vettoretto N, Diaz-Nieto R, Gerych I, Trana C, Faro MP, Yuan KC, Kok KY, Mefire AC, Lee JG, Hong SK, Ghnnam W, Siribumrungwong B, Sato N, Murata K, Irahara T, Coccolini F, Segovia Lohse HA, Verni A, Shoko T. 2013 WSES guidelines for management of intra-abdominal infections. World J Emerg Surg. 2013 Jan 8;8(1):3. doi: 10.1186/1749-7922-8-3. PMID 23294512